CLINICAL TRIAL: NCT02511795
Title: A Phase Ib Study of AZD1775 and Olaparib in Patients With Refractory Solid Tumours
Brief Title: AZD1775 Combined With Olaparib in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6010C00005; REFMAL 384 (Other: Sarah Cannon Development Innovations, LLC)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Refractory Solid Tumours; Relapsed Small Cell Lung Cancer (SCLC)
Keywords: AZD1775; Olaparib; AZD1775 plus Olaparib; Refractory Solid Tumours; Small Cell Lung Cancer (SCLC); Relapsed Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — adavosertib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1775 (6 doses/week) + Olaparib (Experimental): In this Arm, AZD1775 will be given twice daily over 3 days (6 doses) on Days 1-3 of Week 1 and Days 8-10 of Week 2. Olaparib will be given orally BID on Days 1-14.
  All patients will enter an olaparib sub-study in order to assess multiple dose pharmacokinetics of olaparib prior to entering the main study. In the olaparib PK sub-study patients will take olaparib for 3 consecutive days and venous blood samples will be collected on Day 3. The PK sub-study must be initiated 10 days prior to the Cycle 1 Day 1 administration of the AZD1775 and olaparib combination. The patient will experience a short gap in treatment (approximately 4-5 days) between Day 3 of the olaparib PK sub-study and Cycle 1 Day 1 AZD1775 and olaparib combined dosing.
  Interventions: Drug: AZD1775; Drug: Olaparib
- AZD1775 (10 doses/week) + Olaparib (Experimental): In this Arm, AZD1775 will be given twice daily over 5 days (10 doses) on Days 1-5 of Week 1 and Days 8-12 of Week 2. Olaparib will be given orally BID on Days 1-14.
  All patients will enter an olaparib sub-study in order to assess multiple dose pharmacokinetics of olaparib prior to entering the main study. In the olaparib PK sub-study patients will take olaparib for 3 consecutive days and venous blood samples will be collected on Day 3. The PK sub-study must be initiated 10 days prior to the Cycle 1 Day 1 administration of the AZD1775 and olaparib combination. The patient will experience a short gap in treatment (approximately 4-5 days) between Day 3 of the olaparib PK sub-study and Cycle 1 Day 1 AZD1775 and olaparib combined dosing.
  Interventions: Drug: AZD1775; Drug: Olaparib

INTERVENTIONS:
Drug: AZD1775 — AZD1775 will be given twice daily (PO BID) over 3 days (6 doses) on Days 1-3 and 8-10 of each 21 day cycle combined with olaparib PO BID on Days 1-14 of each 21 day cycle.
  Olaparib will be given orally BID on Days 1-14.
Drug: Olaparib — AZD1775 will be given twice daily (PO BID) over 5 days (10 doses) on Days 1-5 and 8-12 of each 21 day cycle combined with olaparib PO BID on Days 1-14 of each 21 day cycle.
  Olaparib will be given orally BID on Days 1-14.

SUMMARY:
The purpose of this Phase 1b, multi-centre, dose escalation study is to find the maximum tolerated dose (MTD) of AZD1775 combined with olaparib in patients with refractory solid tumours

DETAILED DESCRIPTION:
This is a Phase Ib, multi-centre study of AZD1775 combined with olaparib administered orally in patients with refractory solid tumours, or as combination therapy for relapsed small-cell lung cancer (SCLC). There are 2 parts to the study:

Part A: Dose Escalation Part B: Dose Expansion

In Part A, patients with refractory solid tumours will be assessed for safety, tolerability, and pharmacokinetics (PK) of AZD 1775 when combined with olaparib. Different dose levels will be administered to identify the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D).

The dose expansion part (Part B) will further explore the safety, PK, and preliminary efficacy of the AZD1775 RP2D and dosing schedule for the treatment of patients with SCLC who previously had a confirmed response (either a Complete Response or Partial Response) to first-line platinum therapy and then relapsed. Patients who progressed whilst on platinum-containing therapy (platinum refractory) are not permitted to enter the study..

An olaparib pharmacokinetic (PK) sub-study will precede the combined treatment with AZD1775 and olaparib for all patients in Part A. In the sub-study single agent olaparib will be given orally BID for 3 or 5 consecutive days and venous blood samples will be collected on Day 3 or Day 5 as appropriate for assessment of the multiple dose pharmacokinetics of single agent olaparib. Patients will experience a short gap in treatment (approximately 4-5 days) between Day 3 or Day 5 of the olaparib PK sub-study and Cycle 1 Day 1 of the combination treatment.

Patients will continue to receive treatment with AZD1775 and Olaparib until disease progression, intolerable toxicity, or discontinuation criteria have been met.

ELIGIBILITY:
Inclusion Criteria for All Patients

1. Male and female patients ≥ 18 years of age.
2. Any prior palliative radiation therapy must have been completed at least 7 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
4. Baseline laboratory values within 7 days of study drug(s) initiation:

   • ANC ≥ 1500/μL

   • Haemoglobin (Hgb) ≥10 g/dL without transfusion in the past 28 days

   • Platelets ≥ 100,000/μL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN or ≤ 5 x ULN if known liver metastases.
   * Serum bilirubin within normal limits (WNL) or ≤1.5 x ULN in patients with liver metastases, or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well-documented Gilbert's Syndrome.
   * Serum creatinine ≤1.5 x ULN and creatinine clearance (CrCl) ≥ 51 mL/min
5. Female patients who are not of child-bearing potential, and fertile females of childbearing potential who agree to use two highly effective forms of contraception in combination from 2 weeks prior to study treatment and until 1 month after study treatment discontinuation, are not breastfeeding, and must have a negative serum or urine pregnancy test within 28 days of study treatment and confirmed prior to the start of study treatment on first day of dosing.
6. Male patients should be willing to abstain or use barrier contraception (i.e., condoms with a spermicide) for the duration of the study drug exposure and for 3 months after study treatment discontinuation. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential, unless the male patient is abstaining from sexual intercourse.
7. Predicted life expectancy ≥ 12 weeks.

Inclusion Criteria Specific to Part A

1. Histologically confirmed refractory solid tumour for which there is no known or established treatment available with curative intent, after at least one course of systemic therapy for locally advanced or metastatic disease including chemotherapy, targeted therapy or hormonal therapy.
2. Measurable or non-measurable disease according to RECIST v1.1

Inclusion Criteria Specific to Part B

1. Relapsed small-cell lung cancer (SCLC) (defined as a histologically confirmed diagnosis of SCLC) with advanced disease (recurrent or metastatic).
2. Patients must have a confirmed response (either PR or CR) to first-line platinum therapy and then relapsed after completing that treatment. Patients who progressed whilst on platinum-containing treatment (platinum refractory) are not permitted to enter the study. Prior treatment with immunotherapy is permitted..
3. Has agreed to the collection of archival tumour tissue or recent tumor biopsy sample, if taken for routine clinical purposes at baseline if archival tissue is not available for molecular biomarker analyses.
4. Measurable disease according to RECIST v1.1 criteria.

Exclusion Criteria

1. Prior treatment with a PARP inhibitor.
2. Use of an investigational drug during the past 30 days or 5 half-lives (whichever is longer) prior to 1st dose of study treatment.
3. Use of anti-cancer treatment drug ≤ 21 days or 5 half-lives (whichever is shorter) prior to 1st dose of study treatment. For drugs for which 5 half-lives is ≤ 21 days, a minimum of 10 days between termination of the prior treatment and administration of study treatment is required.
4. Radiotherapy (except for palliative reasons) within ≤ 21 days prior to study treatment.
5. No other anti-cancer therapy (except for palliative local radiotherapy), biological therapy, or other novel agent is permitted while the patient is receiving study medication. Patients on luteinizing hormone-releasing hormone (LHRH) analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the investigator.
6. Major surgical procedures ≤ 28 days of beginning study treatment, or minor surgical procedures ≤ 7 days. Patients must have recovered from any of the effects of any major surgery. No waiting period required following port-a-cath placement.
7. Persistent Grade >1 toxicity from prior cancer therapy (except alopecia or anorexia).
8. Patient has an inability to swallow oral medications. Note: Patients with percutaneous endoscopic gastrostomy (PEG) tube or receiving total parenteral nutrition (TPN) are not eligible.
9. Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases, defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment. Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrolment.
10. Patient has had prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to the olaparib PK sub-study dosing and withheld throughout the study until 2 weeks after the last dose of study drug.
11. The use of sensitive substrates of CYP3A4, such as atorvastatin, simvastatin and lovastatin are prohibited in this study. Co-administration of aprepitant or fosaprepitant during this study is prohibited.
12. Caution should be exercised when inhibitors or substrates of P-glycoprotein (P-gp), substrates of CYP1A2 with a narrow therapeutic range, sensitive substrates of CYP2C19 or CYP2C19 substrates with a narrow therapeutic range are administered with AZD1775.

12. Herbal preparations are not allowed throughout the study, including but not limited to: St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng. Patients should stop using these herbal medications 7 days prior to first dose of study treatment.

13. Any known hypersensitivity or contraindication to the components of the study drug AZD1775 or olaparib.

14. Patients with either previous or current myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of MDS/AML.

15. Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥ Class 2.

* Unstable angina pectoris
* Congestive heart failure
* Acute myocardial infarction
* Conduction abnormality not controlled with pacemaker or medication
* Significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)

  16. AZD1775 should not be given to patients who have a history of Torsades des pointes (TdP) unless all risk factors that contributed to TdP have been corrected.

  17. Mean resting corrected QTc interval using the Fridericia formula [QTcF]) ≥ 470 msec for female patients and ≥ 450 msec for male patients from 3 electrocardiograms (ECGs) performed 2-5 minutes apart at study entry or congenital long QT syndrome. .

  18. Pregnant or breastfeeding.

  19. Serious known active infection at the time of enrolment, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.

  20. Presence of other known active invasive cancers.

  21. Psychological, familial, sociological, or geographical conditions that do not permit compliance with protocol.

  22. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (< 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.

  23. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).

  24. Previous allogeneic bone marrow transplant or non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection will exclude patients from the pharmacogenetic portion of the study. If a patient declines to participate in the optional exploratory pharmacogenetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Part A: The incidence of dose-limiting toxicities (DLTs) | 21 days (Cycle 1 duration)
  The maximum tolerated dose (MTD) of the AZD1775/olaparib combination will be the highest dose level at which less than one-third of patients experience a DLT during Cycle 1. Toxicity will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Part B: The incidence of treatment-emergent adverse events (TEAEs) | Up to 12 months
  Treatment-emergent adverse events will be assessed through reports of clinical events and changes from baseline in vital signs and laboratory parameters.

SECONDARY OUTCOMES:
Part A: The incidence of treatment-emergent adverse events (TEAEs). | Up to 12 months
  Treatment-emergent adverse events will be assessed through reports of clinical events and changes from baseline in vital signs and laboratory parameters.
Part A: Peak plasma concentration (Cmax) of olaparib when given as monotherapy in the olaparib PK sub-study. | Olaparib plasma concentration will be measured on Day 3 or Day 5 of the olaparib PK sub-study pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part A: Area under the plasma concentration versus time curve (AUC) of olaparib when given as monotherapy in the olaparib PK sub-study. | Olaparib plasma concentration will be measured on Day 3 or Day 5 of the olaparib PK sub-study: pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part A: Peak plasma concentration (Cmax) of olaparib when given in combination with AZD 1775. | Olaparib plasma conc. will be measured pre-dose & 1, 2, 4, 6, 8, & 10 hours post-dose on Days 3, 8, 10, & 15 (or Days 5, 8, 12, & 15) of Cycle 1; & Days 1, 3, & 8 (or Days 1, 5, & 8) of Cycle 2; & Days 3 or 10 (or Days 5 or 12) of Cycle 3.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib when given in combination with AZD1775. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part A: Area under the plasma concentration versus time curve (AUC) of olaparib when given in combination with AZD 1775. | AUC for olaparib will be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3, 8, 10, and 15 (or Days 5, 8, 12, and 15) of Cycle 1; and Days 1, 3, and 8 (or Days 1, 5, and 8) of Cycle 2; and Days 3 or 10 (or Days 5 or 12) of Cycle 3.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib when given in combination with AZD1775. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part A: QTc Interval | Pre-dose and at pre-specified times on Day 1 and 3 (or 5) of the olaparib PK sub-study, prespecified times on Days 1, 3, and 10 (or 1, 5, and 12) of Cycle 1, and pre-specified times on Days 1 and 3 (or 1 and 5) of Cycle 2, up to 9 weeks.
  Triplicate 12-lead ECGs will be performed approximately 2-5 minutes apart. The QTc interval will be calculated using Friderica's formula.
Part A: Peak plasma concentration (Cmax) of AZD1775 when given in combination with olaparib. | AZD1775 plasma conc. will be measured pre-dose & 1, 2, 4, 6, 8, & 10 hours post-dose on Days 3, 8, 10, & 15 (or Days 5, 8, 12, & 15) of Cycle 1; & Days 1, 3, & 8 (or Days 1, 5, & 8) of Cycle 2; & Days 3 or 10 (or Days 5 or 12) of Cycle 3.
  Pharmacokinetic parameters will be derived from the plasma concentration data for AZD1775 given in combination with olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part A: Area under the plasma concentration versus time curve (AUC) of AZD1775 when given in combination with olaparib. | AUC for AZD1775 be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3, 8, 10, and 15 (or Days 5, 8, 12, and 15) of Cycle 1; and Days 1, 3, and 8 (or Days 1, 5, and 8) of Cycle 2; and Days 3 or 10 (or Days 5 or 12) of Cycle 3.
  Pharmacokinetic parameters will be derived from the plasma concentration data for AZD1775 when given in combination with olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part B: Peak plasma concentration (Cmax) of olaparib when given in combination with AZD1775. | Olaparib plasma concentration will be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3 and 10 of Cycle 1.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib given in combination with AZD1775. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part B: Area under the plasma concentration versus time curve (AUC) of olaparib when given in combination with AZD1775. | AUC for olaparib will be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3 and 10 of Cycle 1.
  Pharmacokinetic parameters will be derived from the plasma concentration data for olaparib when given in combination with AZD1775. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part B: Peak plasma concentration (Cmax) of AZD1775 when given in combination with olaparib. | AZD1775 plasma concentration will be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3 and 10 of Cycle 1.
  Pharmacokinetic parameters will be derived from the plasma concentration data for AZD1775 given in combination with olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part B: Area under the plasma concentration versus time curve (AUC) of AZD1775 when given in combination with olaparib. | AUC for AZD1775 will be measured pre-dose and 1, 2, 4, 6, 8, and 10 hours post-dose on Days 3 and 10 of Cycle 1.
  Pharmacokinetic parameters will be derived from the plasma concentration data for AZD1775 when given in combination with olaparib. The date and actual time of the PK sample is to be recorded in the medical records and eCRF.
Part B: Presence of genetic alterations | Screening (prior to any study treatment), or at any visit throughout the life of the study (up to approximately 12 months).
  If the patient has given informed consent for genetic sampling and analysis a 10 mL sample of whole blood will be collected and tested for the presence of genetic alterations.
Objective Response Rate (ORR) | Through study completion (an average of 6 months)
  The objective response rate (ORR) is the number of patients with a confirmed best objective response of Complete Response (CR) or Partial Response (PR) divided by the number of patients in the full analysis set with measurable disease at baseline. ORR is determined by the Investigator in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Progression-Free Survival (PFS) | From the beginning of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival (PFS) is defined as the time from the beginning of treatment to disease progression or death from any cause.
Overall Survival (OS) | From the beginning of treatment until the date of death from any cause, assessed up to 12 months.
  Overall survival (OS) is defined as the time from the beginning of treatment to death from any cause.
Disease Control Rate (DCR) | Through study completion (an average of 6 months)
  Disease Control Rate (DCR) is defined (RECIST v1.1) as the percentage of patients in the full analysis set with a confirmed best objective response of complete response (CR), partial response (PR), or a best objective response of stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Erika P. Hamilton, M.D., Principal Investigator — SCRI Development Innovations, LLC
Locations (6):
- United States (5):
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Research Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton EP, Falchook GS, Wang JS, Fu S, Oza AM, Imedio ER, Kumar S, Ottesen L, Mugundu GM, de Bruin EC, O'Connor MJ, Jones SF, Spigel DR, Li BT. Adavosertib in Combination with Olaparib in Patients with Refractory Solid Tumors: An Open-Label, Dose-Finding, and Dose-Expansion Phase Ib Trial. Target Oncol. 2024 Nov;19(6):879-892. doi: 10.1007/s11523-024-01102-8. Epub 2024 Nov 1. PMID 39487373